CLINICAL TRIAL: NCT05471921
Title: Effectiveness of an Evidence-based Stepped Care System for Alcohol and Other Drug Use Problems Among Congolese Refugees in Zambia: A Randomized Controlled Trial
Brief Title: Effectiveness of an Evidence-based Stepped Care System for Alcohol and Other Drug Use Problems Among Congolese Refugees in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Elrha (Other)
Responsible Party: Principal Investigator, Jeremy C. Kane, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU0532
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Alcohol and Substance-Related Mental Disorders
Keywords: Alcohol Use Disorder; Substance Use Disorders; Depression; Anxiety; Trauma
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Depression; Anxiety Disorders; Wounds and Injuries | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized to SBIRT or treatment as usual (TAU) control. The Research Assistant (RA) will allocate participants to study conditions using a series of sealed, opaque envelopes. RAs and data analysts will be blinded. Participants will be notified immediately about the result of the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBIRT (Experimental): Experimental condition: Participants residing in the study community (displaced and host population) will receive Screening, Brief Intervention, and Referral to Treatment (SBIRT). The treatment will consist of brief intervention (CETA-BI) and full Common Elements Treatment Approach (CETA) depending on the severity of the participant's substance use.
  Interventions: Behavioral: SBIRT
- Treatment as usual (Active Comparator): Comparison condition: Participants residing in the study community (displaced and host population) will receive the current standard of treatment.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: SBIRT — SBIRT is an evidence-based treatment for unhealthy alcohol and other drugs (AOD) use in non-humanitarian settings and can efficiently provide individuals with an appropriate level of care based on their symptoms. Participants randomized to SBIRT will receive an on-the-spot alcohol brief intervention (CETA-BI) and be categorized as low or moderate/high severity using the AUDIT scale. Participants who are moderate/high severity will be connected to a counselor and will begin full CETA treatment. CETA is a transdiagnostic approach that combines motivational interviewing with cognitive behavioral therapy to assist clients in considering changing their rates of AOD use. The intervention lasts 30-40 minutes and consists of 6 components including 1) screening; 2) identifying the impacts of unhealthy AOD use; 3) talking about change/goal-setting; 4) understanding the primary reason for drinking; 5) skill-building; and 6) referral for services.
  Arms: SBIRT
Behavioral: Treatment as usual — Mantapala health workers and supervisors were trained in mental health gap action program-humanitarian intervention guide (mhGAP-HIG), which is a mental health service provision guide for use in humanitarian settings; this training was led by staff from United Nations High Commissioner for Refugees. This training did not include evidence-based psychological interventions (e.g., CETA). Participants randomized to TAU will be referred to the existing services that exist in the health clinic located in Mantapala refugee settlement. More specialized services are referred to the District Hospital in Nchelenge.
  Arms: Treatment as usual

SUMMARY:
This is a randomized controlled trial (RCT) evaluating the effectiveness of a screening, brief intervention, and referral to treatment (SBIRT) stepped-care system in reducing unhealthy AOD use among Congolese refugees and the host community in Mantapala, an integrated settlement in northern Zambia.

DETAILED DESCRIPTION:
Refugees are at risk for unhealthy alcohol and other drug (AOD) use, particularly in protracted emergencies. The investigators define unhealthy AOD use as hazardous use, harmful use, and alcohol/substance use disorder and dependence. Among refugees, baseline risk for AOD use may increase for several reasons, including access to illicit substances (reduced drug enforcement policies and security), exposure to potentially traumatic events, and chronic adversity. Ongoing adverse environments such as refugee camps, are associated with lack of access to basic needs, limited livelihoods opportunities, boredom, marginalization, loss of resources, and mental health problems leading to the use of AOD as a coping mechanism. Studies have suggested that in conflict settings, quantity and frequency of use tend to increase from the pre-conflict stage to peri- and post-conflict. Increase in use of one substance can also lead to initiation of new substances, resulting in more complex cases of polysubstance use.

In Mantapala refugee settlement in Zambia, the proposed study setting, unhealthy AOD use is reportedly common. In July 2019, United Nations High Commissioner for Refugees (UNHCR) requested psychiatric clinical officers from local health facilities in Nchelenge, Zambia to do an assessment of mental health problems among refugees in Mantapala. The community-based convenience sample consisted of 200 people, of whom 35 (18%) had probable alcohol use disorder, mostly adult men and adolescents (male and female), and frequent cannabis use among people who were drinking alcohol. Reports from 7 refugee incentive workers and 17 representatives from 6 implementing agencies during an initial site visit indicated that unhealthy AOD use was associated with individual, family, and community consequences (injury, gender-based violence, diversion of livelihoods). Reports from the province of origin (Katanga, DRC) and host country (Zambia) have also found AOD use to be prevalent.

The proposed study will test an intervention package known as 'screening, brief intervention, and referral to treatment' (SBIRT). SBIRT systems are evidence-based for the treatment of unhealthy AOD use in non-humanitarian settings and can efficiently provide individuals with an appropriate level of care based on their symptom presentation and severity. For example, individuals with hazardous AOD use but without a more severe disorder and without mental health comorbidities may be best served by a brief intervention (BI); for many of these individuals, a full course of a psychotherapy may not be necessary (i.e., inefficient use of limited resources). On the other hand, individuals with more severe AOD disorder or mental health comorbidities likely require more comprehensive treatment. In this trial the investigators will provide BI or BI+psychotherapy commensurate with an individual's symptom presentation.

The interventions included in the SBIRT system are the Common Elements Treatment Approach-Brief Intervention (CETA-BI) and the full CETA psychotherapy (CETA). Previous randomized controlled trials have found CETA to be an effective treatment, including among refugees, for a range of mental and behavioral health problems, including depression, anxiety, trauma, and functional impairment. CETA has recently been tested in Zambia and found to also reduce unhealthy alcohol use in addition to mental health problems and intimate partner violence. CETA is a transdiagnostic approach, meaning that counselors trained in CETA are equipped with the ability to treat a range of co-occurring mental and behavioral health conditions. It was developed for use in low- and middle-income countries (LMIC) to facilitate lower cost and sustainability. CETA includes 9 cognitive behavioral elements found in most evidence-based psychological treatments. CETA is 6-12 weekly one-hour sessions with flexibility depending on symptom severity. CETA-BI combines motivational interviewing skills with cognitive behavioral therapy to assist clients in considering changing their rates of AOD use. The intervention lasts 30-40 minutes and consists of 6 components including: 1) screening; 2) identifying the impacts of unhealthy AOD use; 3) talking about change and goal-setting; 4) understanding the primary reason for drinking; 5) skill building; and 6) referral for services. CETA-BI and CETA were previously found effective for AOD use and mental health problems within HIV care in Lusaka, Zambia. CETA-BI and CETA have significant potential for adaptation and implementation in refugee settings but a rigorous RCT adapting and testing them in an SBIRT stepped-care approach among refugees is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Living in Mantapala refugee settlement (i.e., Congolese refugee) or (Zambian) member of neighboring host community
* Unhealthy alcohol use based on standard cut-off scores of the ACASI-based Alcohol Use Disorders Identification Test (AUDIT)20 (≥ 8 for men and ≥ 4 for women).21 The focus on unhealthy alcohol use as the primary inclusion criterion is due to preliminary research in Mantapala suggesting that alcohol is the main substance of concern and other drug use almost exclusively co-occurs with alcohol use.

Exclusion Criteria:

* Severe psychiatric illness, high suicide risk (based on recent attempts and/or ideation with intent and plan), and/or current severe AOD withdrawal that would necessitate immediate referral for psychiatric services
* Inability or unwillingness to provide informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Kane, PhD, Principal Investigator — Columbia University; Claire Greene, PhD, Principal Investigator — Columbia University; Muzi Kamanga, Principal Investigator — Women in Law and Development in Africa (WiLDAF); Henry Loongo, PhD, Principal Investigator — CARE Zambia
Locations (2):
- Columbia University, New York, New York, United States
- Mantapala Refugee Settlement, Nchelenge, Luapula Province, Zambia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SBIRT | Treatment as usual
Started | 199 | 201
Completed | 157 | 153
Not Completed | 42 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBIRT | Treatment as usual | Total
Number analyzed (Participants) | 199 | 201 | 400
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.8 (12.3) | 36.9 (11.9) | 36.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 58 | 113
  Male | 144 | 143 | 287
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 199 | 201 | 400
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Nationality [Count of Participants; unit: Participants]
  Congolese | 115 | 117 | 232
  Zambian | 84 | 84 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change in Alcohol Use Disorders Identification Test (AUDIT) Score
Description: AUDIT is a 10-item measure of hazardous alcohol use with a possible range of 0-40 (total scale score). Higher scores are associated with more hazardous use.
Time Frame: Baseline, 6-months, 12-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT | Treatment as usual
Number analyzed (Participants) | 199 | 201
score on a scale
  Mean change from Baseline to 6 months | -12.6 [-14.3 to -11.0] | -8.1 [-9.8 to -6.3]
  Mean change from Baseline to 12 months | -13.8 [-15.5 to -12.1] | -10.3 [-12.1 to -8.6]

2. Secondary Outcome: Change in Center for Epidemiologic Studies - Depression Scale (CES-D) Score
Description: The CES-D is a is a 20-item measure that asks individuals to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Time Frame: Baseline, 6-months, 12-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT | Treatment as usual
Number analyzed (Participants) | 199 | 201
score on a scale
  Mean change from Baseline to 6 months | -9.5 [-11.6 to -7.5] | -5.8 [-7.9 to -3.7]
  Mean change from Baseline to 12 months | -8.9 [-11.0 to -6.8] | -8.1 [-10.3 to -6.0]

3. Secondary Outcome: Change in Generalized Anxiety Disorder-7 Scale (GAD-7) Score
Description: The GAD-7 questionnaire is a seven-item, self-report anxiety questionnaire designed to assess the patient's health status. Scores of 0, 1 or 2 are given for experiencing symptoms 'not at all', for 'several days', for 'more than half the days' and for 'nearly every day', respectively. The scores are then totaled and presented from 0 to 21, with high scores indicating greater anxiety symptoms.
Time Frame: Baseline, 6-months, 12-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT | Treatment as usual
Number analyzed (Participants) | 199 | 201
score on a scale
  Mean change from Baseline to 6 months | -3.6 [-4.5 to -2.6] | -2.1 [-3.0 to -1.2]
  Mean change from Baseline to 12 months | -3.5 [-4.4 to -2.6] | -3.2 [-4.1 to -2.2]

4. Secondary Outcome: Change in Harvard Trauma Questionnaire (HTQ)
Description: HTQ is a checklist that inquires about a variety of trauma events, as well as the emotional symptoms considered to be uniquely associated with trauma. The HTQ is a 39-item PTSD symptom scale with a possible range of 1-4 (average scale score). Higher scores are associated with greater PTSD symptom severity.
Time Frame: Baseline, 6-months, 12-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT | Treatment as usual
Number analyzed (Participants) | 199 | 201
score on a scale
  Mean change from Baseline to 6 months | -0.5 [-0.6 to -0.4] | -0.4 [-0.5 to -0.3]
  Baseline to 12 months | -0.5 [-0.6 to -0.4] | -0.5 [-0.6 to -0.4]

5. Secondary Outcome: Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST): Risk Score (Continuous Outcome)
Description: The ASSIST is a questionnaire that screens for all levels of problem or risky substance use in adults. The ASSIST consists of eight questions covering tobacco, alcohol, cannabis, cocaine, amphetamine-type stimulants (including ecstasy) inhalants, sedatives, hallucinogens, opioids and 'other drugs'. A risk score is provided for each substance, and a total risk score is calculated with a minimum score of 0 and a maximum score of 243. Higher scores are indicative of higher risk substance use.
Time Frame: Baseline, 6-months, 12-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SBIRT | Treatment as usual
Number analyzed (Participants) | 199 | 201
score on a scale
  Mean change from baseline to 6 months | -28.3 [-34.7 to -21.8] | -23.0 [-29.5 to -16.4]
  Mean change from baseline to 12 months | -30.4 [-36.9 to -24.0] | -26.1 [-32.6 to -19.5]

6. Secondary Outcome: Number of Participants Who Had Any Substance Use in the Past 3 Months, Based on Responses to the ASSIST Questionnaire
Description: as for outcome 5
Time Frame: Baseline, 6-months, 12-months
Measure: Count of Participants; unit: Participants
Arm/Group | SBIRT | Treatment as usual
Number analyzed (Participants) | 199 | 201
Participants
  Baseline | 60 | 55
  6 months | 24 | 33
  12 months | 18 | 22

7. Secondary Outcome: Sleep Scale for the Medical Outcomes Research Study
Description: The Medical Outcomes Study Sleep Scale includes 12 items assessing sleep disturbance, sleep adequacy, somnolence, quantity of sleep, snoring, and awakening short of breath or with a headache. The scores of the dimensions and of the sleep problem index were converted to a 0 to 100 scale, with higher scores reflecting more of the attribute implied by the name (e.g. greater sleep disturbance, greater adequacy of sleep).
Time Frame: Baseline, 6-months, 12-months
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | SBIRT | Treatment as usual
All-Cause Mortality (participants affected / at risk) | 0/199 | 3/201
Serious Adverse Events (participants affected / at risk) | 8/199 | 1/201
Other Adverse Events (participants affected / at risk) | 0/199 | 0/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBIRT (N=199) | Treatment as usual (N=201)
Hospitalization (Infections and infestations) | 4 (4) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Intimate partner violence (Social circumstances) | 1 (1) | 0 (0)
Hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0)
Illness (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT05471921/Prot_SAP_000.pdf